CLINICAL TRIAL: NCT07051148
Title: Efficacy of a Personalized, Response-based Transdiagnostic Intervention for Emotional Disorders Delivered Via the Internet: A Protocol for an Adaptive Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Jaume I (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TRANSBLEND
Record Dates: First submitted 2025-05-26; First posted 2025-07-03 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Emotional Disorders; Anxiety; Depression, Unipolar
Keywords: transdiagnostic; internet based therapy; anxiety; depression; Emotional Disorders; adaptive intervention; blended treatment; digital interventions; personalization; personalized treatment; adaptive trial
MeSH Terms: conditions — Anxiety Disorders; Depressive Disorder; Depression

STUDY DESIGN:
Intervention Model Description: Multivarate experimental adaptive design (2 factors, 4 groups). Randomization will occur after the initial intervention phase (first 3 modules), based on symptom reduction using a Reliable Change Index (RCI). Participants will be classified as early or late responders. Within each group, simple randomization (1:1) will be implemented using a computer-generated sequence (in R). Assignment will be managed by and external researcher blind to clinical staff, using preloaded, password-protected lists. No stratification by sex, age or sociocultural status will be applied.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Early responders selfapplied completed (Experimental)
  Interventions: Behavioral: UJI Online Transdiagnostic Protocol
- Early responders selfapplied interrupted (Experimental)
  Interventions: Behavioral: UJI Online Transdiagnostic Protocol
- Late responders selfapplied (Experimental)
  Interventions: Behavioral: UJI Online Transdiagnostic Protocol
- Late responders blended (Experimental)
  Interventions: Behavioral: UJI On Line Transdiagnostic Hibrid Protocol

INTERVENTIONS:
Behavioral: UJI Online Transdiagnostic Protocol — Is a manualized treatment for emotional disorders delivered through an interactive multimedia platform. The self applied format consists of 12 self applied modules (psychoeducation, emotional processing, cognitive flexibility training, exposure, coping strategies, maladaptive behaviors, avoidance, etc)
  Arms: Early responders selfapplied completed; Early responders selfapplied interrupted; Late responders selfapplied
Behavioral: UJI On Line Transdiagnostic Hibrid Protocol — Hybrid format: 12 self applied modules with two synchronous sessions with a trained therapist
  Arms: Late responders blended

SUMMARY:
This adaptive randomized controlled trial evaluates the efficacy of a transdiagnostic, internet-delivered psychological intervention for emotional disorders, tailored to patient´s early clinical response. 366 adults with clinically significant symptoms of depression and/or anxiety will begin a 12 module self-applied program. Based on sympron reduction after the first three modules, participants will be classified as early or late responders and randomized into different experimental arms. The main hypothesis is that a hybrid format (self-applied modules plus synchronous sessions with a therapist) will yield better outcomes for late responders. Outcomes include symptom reduction, emotional regulation and internet based therapheutic alliance.

DETAILED DESCRIPTION:
To assess its effectiveness, two formats will be compared: the original, consisting of 12 self-administered modules, and a hybrid format, which includes two synchronous sessions with a trained therapist. Early responders will either continue with the original intervention or discontinue treatment; while late responders will receive the hybrid format or continue with the original intervention. The primary expected result is that the hybrid format will improve treatment outcomes for late responders compared to the self-applied format. The findings are expected to inform clinical practice by highlighting the importance of assessing symptomatic response throughout treatment, especially in its early phases

ELIGIBILITY:
Inclusion Criteria:

* Spanish speakers
* PHQ 9 score + 5
* GAD 7 score + 5
* Access to Internet
* Email

Exclusion Criteria:

* Severe mental disorder: schizophrenia/bipolar disorder
* Active substance abuse
* High suicide risk
* Ongoing psychological/pharmacological treatment
* Interfering physical illness

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 366 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Clinical Outcomes in Routine Evaluation (CORE-34, Evans et al., 2002) | Day 1 Week 1, 2, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13 Week 25 Year 1
  Is a self report questionnaire designed to assess psychological distress and global functioning across four domains: subjective well being, problems/symptoms, functioning and risk. Items are rated on a 5 point Likert scale. The instrument has demostrated good psychometrics properties. Higher scores indicate greater psychological distress.
Patient Health Questionnaire (PHQ-9; Kroenke et al., 2001) | Day 1 Week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13 Week 25 Year 1
  Is a 9 item self report scale used to asses the severity of depressive symptoms over the past two weeks. Items are rated on a 4 point Likert scale (0-3). Is widely used in clinical and research settings, with strong psychometric properties of reliability and validity.
Generalized Anxiety Disorder scale (GAD-7, Spitzer et al., 2006) | Day 1 Week 1, 2, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13 Week 25 1 Year
  Is a 7 item self report questionnaire designed to asses the severity to generalized anxiety symptoms over the past two weeks. Items are rated in a 4 point Likert scale (0-3). Is widely used in clinical and research settings, with strong psychometrics properties of reliability and validity.

SECONDARY OUTCOMES:
State Difficulties in Emotion Regulation Scale (S-DERS, Lavender et al., 2017) | Day 1 Week 4, 8, 13 Week 25 Year 1
  Is a 21 item self report scale that asseses momentary difficulties in emotion regulation across 4 domains: nonacceptance, modulation, awareness and clarity. Respondents rate their emotional experience in a 5 points Likert scale. The instrument is sensitive to short term fluctuations and is suitable for evaluating changes in emotion regulation during treatment.
Inventory of Interpersonal Problems (IIP32, Horowitz, 2000) | Day 1 Week 4, 8, 13 Week 25 Year 1
  Is is a self-report questionnaire designed to assess interpersonal difficulties experienced over the past month. It covers eight dimensions of interpersonal functioning (e.g., being too controlling, socially inhibited, or self-sacrificing). Each item is rated on a 5-point Likert scale. The IIP-32 is a widely validated and efficient tool for identifying interpersonal patterns relevant to psychological distress and treatment planning.

OTHER OUTCOMES:
Working Alliance Inventory for Internet Interventions (WAI-I; Gómez Penedo et al., 2020) | Day 1 Week 4, 8, 13
  Is a 12-item self-report measure adapted from the traditional Working Alliance Inventory to assess the therapeutic alliance in the context of internet-based psychological interventions. It evaluates three core dimensions: agreement on tasks, agreement on goals, and the bond between the patient and the program or supporting professional. Items are rated on a 5-point Likert scale. The WAI-I has demonstrated good psychometric properties in online intervention settings.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://doi.org/10.1007/978-3-319-91776-4_4
- See also: Related Info — https://preprints.jmir.org/preprint/45135
- See also: Related Info — https://doi.org/10.2147/NDT.S93315
- See also: Related Info — https://doi.org/10.1016/j.invent.2023.100670
- See also: Related Info — https://doi.org/10.1146/annurev-clinpsy-080822-051119
- See also: Related Info — https://doi.org/10.1186/s12888-017-1297-z
- See also: Related Info — https://doi.org/10.2196/jmir.6588
- See also: Related Info — https://doi.org/10.1016/j.invent.2024.100715
- See also: Related Info — https://doi.org/10.1016/j.cpr.2019.101810
- See also: Related Info — https://doi.org/10.1016/j.invent.2023.100601